CLINICAL TRIAL: NCT04902508
Title: Evaluation of an Explicit Approach to Teach Grammatical Forms to Children With Language Impairment
Brief Title: Evaluation of an Explicit Approach
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: R01DC019374-01 (NIH)
Record Dates: First submitted 2021-05-17; First posted 2021-05-26 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Developmental Language Disorder; Explicit Intervention; Grammatical Language
Keywords: Child Language; Randomized Control Trial; Intervention; Grammar; Morphology
MeSH Terms: conditions — Language Development Disorders

STUDY DESIGN:
Intervention Model Description: This study uses a sequential multiple assignment randomized trial (SMART) design with two phases of randomization.
Who Masked: Investigator, Outcomes Assessor
Masking Description: All assessors will be blinded to intervention assignments. To reduce assessor bias, after Phases 1 and 2, two different trained research assistants unfamiliar with the participant will administer the Grammatical Language Probe. These same examiners may administer the 1-, 6-, and 12-month assessments. The PIs and board of advisors will also be blinded to intervention assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Explicit Master Plus No Additional Treatment (Experimental): Receives 32 sessions of explicit treatment then assessed. When assessed, demonstrates "Mastery" and receives no additional treatment.
  Interventions: Behavioral: Explicit-added
- Explicit Master Plus Explicit Treatment (Experimental): Receives 32 sessions of explicit treatment then assessed. When assessed, demonstrates "Mastery" and receives 32 additional sessions of explicit treatment.
  Interventions: Behavioral: Explicit-added
- Explicit Master Plus Implicit Treatment (Experimental): Receives 32 sessions of explicit treatment then assessed. When assessed, demonstrates "Mastery" and receives 32 sessions of implicit treatment.
  Interventions: Behavioral: Implicit-only; Behavioral: Explicit-added
- Explicit Non-Master Plus Explicit Treatment (Experimental): Receives 32 sessions of explicit treatment then assessed. When assessed, demonstrates "Non-Mastery" and receives 32 additional sessions of explicit treatment.
  Interventions: Behavioral: Explicit-added
- Explicit Non-Master Plus Implicit Treatment (Experimental): Receives 32 sessions of explicit treatment then assessed. When assessed, demonstrates "Non-Mastery" and receives 32 sessions of implicit treatment.
  Interventions: Behavioral: Implicit-only; Behavioral: Explicit-added
- Implicit Master Plus No Additional Treatment (Experimental): Receives 32 sessions of implicit treatment then assessed. When assessed, demonstrates "Mastery" and receives no additional treatment.
  Interventions: Behavioral: Implicit-only
- Implicit Master Plus Implicit Treatment (Experimental): Receives 32 sessions of implicit treatment then assessed. When assessed, demonstrates "Mastery" and receives 32 additional sessions of implicit treatment.
  Interventions: Behavioral: Implicit-only
- Implicit Master Plus Explicit Treatment (Experimental): Receives 32 sessions of implicit treatment then assessed. When assessed, demonstrates "Mastery" and receives 32 sessions of explicit treatment.
  Interventions: Behavioral: Implicit-only; Behavioral: Explicit-added
- Implicit Non-Master Plus Implicit Treatment (Experimental): Receives 32 sessions of implicit treatment then assessed. When assessed, demonstrates "Non-Mastery" and receives 32 additional sessions of implicit treatment.
  Interventions: Behavioral: Implicit-only
- Implicit Non-Master Plus Explicit Treatment (Experimental): Receives 32 sessions of implicit treatment then assessed. When assessed, demonstrates "Non-Mastery" and receives 32 sessions of explicit treatment.
  Interventions: Behavioral: Implicit-only; Behavioral: Explicit-added

INTERVENTIONS:
Behavioral: Implicit-only — Each intervention session will comprise four core activities: sentence imitation, presentation of a model story with production opportunities, and auditory bombardment.
  Arms: Explicit Master Plus Implicit Treatment; Explicit Non-Master Plus Implicit Treatment; Implicit Master Plus Explicit Treatment; Implicit Master Plus Implicit Treatment; Implicit Master Plus No Additional Treatment; Implicit Non-Master Plus Explicit Treatment; Implicit Non-Master Plus Implicit Treatment
Behavioral: Explicit-added — Each intervention session will comprise four core activities: sentence imitation, presentation of a model story with production opportunities, and auditory bombardment. Interventionists will also present the rule/pattern guiding the target form.
  Arms: Explicit Master Plus Explicit Treatment; Explicit Master Plus Implicit Treatment; Explicit Master Plus No Additional Treatment; Explicit Non-Master Plus Explicit Treatment; Explicit Non-Master Plus Implicit Treatment; Implicit Master Plus Explicit Treatment; Implicit Non-Master Plus Explicit Treatment

SUMMARY:
This study is a randomized clinical trial that uses a Sequential Multiple Assignment Randomized Trial (SMART) study design. The study will directly compare the efficacy of an innovative intervention that combines explicit and implicit approaches to a traditional implicit treatment approach to teach true grammatical forms to children with developmental language disorder (DLD). The study will also compare interventions that include sequences of Explicit-added and Implicit-only treatments. Participants will include 5- through 9-year-old children with DLD who present with significant grammatical weaknesses. In Phase 1, 155 participants will be randomized 1:1 to an Explicit-added treatment group or an Implicit-only treatment group. Each participant will complete 32 sessions targeting four unique grammatical forms (8 sessions/form). In Phase 2, "Masters" will be re-randomized to receive no treatment 32 sessions of the same treatment, or 32 sessions of the alternative treatment. "Non-Masters" will be re-randomized to receive 32 additional sessions of the same treatment or 32 sessions of the alternative treatment. Performance will be measured on acquisition, maintenance, and generalization probes obtained immediately,1-, 6-, and 12- months post-intervention. The SMART study design will be used to determine if child factors, including expressive and receptive language abilities, nonverbal IQ, and executive function skills can reliably predict the treatment sequence that optimizes language learning. Study results will help to determine the best sequence approach to ameliorate grammatical weaknesses, one of the core deficits of young children with language impairment.

DETAILED DESCRIPTION:
This study is a randomized trial with two phases. Phase 1 is a traditional randomized trial during which eligible and consenting participants will be randomized equally to one of two interventions: Explicit-added or Implicit-only. Randomization is blocked by age (5- & 6-year-olds; and 7- to 9-year-olds) and receptive language ability to ensure that ages are matched across groups and that half of the participants in each treatment group have receptive language skills below average. A standard score of 80 is used to categorize participants (below average: < 80; average: ≥ 80) based on the Receptive Language Index of the Clinical Evaluation of Language Fundamentals (CELF). Participants are also stratified based on child gender. All participants will complete 32 sessions (8 sessions per target in blocks of 4). In Phase 2, participants in both the Explicit-added and Implicit-only groups will be re-randomized based on level of mastery on treatment goals. Participants who are considered treatment "Masters" and have achieved the criterion of 80% accuracy on all target forms will be re-randomized to receive no further treatment or a round of the alternative treatment. Participants who have not yet mastered each of the four target forms (< 80% accuracy) will be re-randomized to receive another round of either the same treatment or the alternative treatment.

Study participants will include 155 children with language impairment, aged 5 through 9 years, accounting for a 10% attrition rate resulting in 140 participants. This age includes children who likely experience difficulties with the grammatical forms targeted in intervention and who are receiving intervention for weaknesses in grammatical language. Researchers will recruit participants with an effort to maximize participant diversity based on ethnicity and parental education. We aim to recruit a representative sample of children with DLD, which will include more boys than girls. Participants will not have any indication of other significant conditions to which their impairment may be attributed, such as autism spectrum disorder, Down syndrome, seizure disorder, or hearing impairment. Participants with a diagnosis of attention deficit/hyperactivity disorder will be included due to high rate of co-morbidity.

ELIGIBILITY:
Inclusion Criteria:

Study participants will include children with language impairment, aged 5 through 9 years. Participants will not have any indication of other significant conditions to which their impairment may be attributed, such as autism spectrum disorder, Down syndrome, seizure disorder, or hearing impairment. Participants with a diagnosis of attention deficit/hyperactivity disorder will be included due to high rate of co-morbidity (see Redmond, 2016). Additionally, participants will meet the following criteria:

* No evidence of significant cognitive delay;
* Evidence of language impairment;
* Evidence of deficits on expressive grammatical forms: score below 30% accuracy on at least two of the following forms: third person singular -s, regular past tense -ed, auxiliary is/are in statements, auxiliary do/does in questions;
* Typical hearing and vision, with correction if necessary;
* Native English speaker with English spoken in the home by at least one primary caregiver since birth;
* Speaker of Mainstream American English;
* Be able to articulate final-position phonemes /s/, /z/, /t/, and /d/; and
* Majority of utterances (> 50%) include subject and verb in obligated contexts based on a 20-min conversational language sample to ensure appropriateness of study intervention.

Exclusion Criteria:

Participants will be excluded if there is no indication of language impairment, and they are not aged 5 through 9 years. Participants will also be excluded if there is indication of other significant conditions to which their impairment may be attributed, such as autism spectrum disorder, Down syndrome, seizure disorder, or hearing impairment. Additionally, participants will be excluded in they meet the following criteria:

* Evidence of significant cognitive delay;
* No evidence of deficits on expressive grammatical forms: score below 30% accuracy on at least two of the following forms: third person singular -s, regular past tense -ed, auxiliary is/are in statements, auxiliary do/does in questions;
* Atypical hearing and vision, with correction if necessary;
* Non-native English speaker;
* Speaker of Non-mainstream American English;
* Unable to articulate final-position phonemes /s/, /z/, /t/, and /d/; and
* Non-majority of utterances (< 50%) include subject and verb in obligated contexts based on a 20-min conversational language sample to ensure appropriateness of study intervention.

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 111 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Grammatical Language Probe | After 32 sessions or approximately 4 months.
  The primary outcome measure will be the change in percentage correct on the Grammatical Language Probe from pre- to post-intervention. The researcher-developed 64-item probe contains 8 contrastive pairs of each of the four target forms. Half of the verbs used in the sentence pairs will comprise verbs intentionally included in session models and recasts; half will include verbs not intentionally included in models and recasts. Participants will be shown a picture and prompted to describe the picture using the target form. Scores will range from 0-64, with higher indicating better performance. Percent correct will be used in analyses.

SECONDARY OUTCOMES:
Structured Photographic Picture Language Test - 3 (SPELT-3) | After 64 sessions (or approximately 8 months) and 6-months, and 12-months post intervention
  The SPELT-3 includes 54 full color photographs of everyday situations and objects paired with simple verbal questions and statements to elicit 22 morphological and syntactic structures. Standard scores (mean = 100; SD = 15) will be used in analyses.
Mean Length of Utterance - Morphemes (MLU-m) | After 64 sessions (or approximately 8 months) and 6-months, and 12-months post intervention
  The MLU-m will be derived from a 20-min language sample with a researcher. MLU-m may range from 0 and on. Higher MLU-m typically reflects greater sentence complexity. MLU-m will be used in study analyses.
Developmental Sentence Scoring (DSS) | After 64 sessions (or approximately 8 months) and 6-months, and 12-months post intervention
  The DSS will be derived from a 20-min language sample with a researcher. The DSS may range from 0 to 8. Higher DSS scores typically reflects greater sentence complexity. The average DSS will be used in study analyses.
Grammatical Language Probe | After 64 sessions (or approximately 8 months) and 6-months, and 12-months post intervention
  The primary outcome measure will be the change in percentage correct on the Grammatical Language Probe. The researcher-developed 64-item probe contains 8 contrastive pairs of each of the four target forms. Half of the verbs used in the sentence pairs will comprise verbs intentionally included in session models and recasts; half will include verbs not intentionally included in models and recasts. Participants will be shown a picture and prompted to describe the picture using the target form. Scores will range from 0-64, with higher indicating better performance. Percent correct will be used in analyses.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
Only de-identified data will be shared. Identifying information will be stripped and kept confidential. Data that will be stored includes performance raw and standard scores on all assessments and de-identified written transcripts of language samples obtained. Participants will be given information regarding data sharing and will consent to data sharing.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Five years after publication of the last manuscript de-identified data will be made available online via the lab website or other public data repository. Non-identifying scripts and descriptions of data analysis techniques will be made public immediately upon publication through the same methods.
Access Criteria: De-identified data, metadata, and analysis information will be shared publicly online. Access will not be restricted.